CLINICAL TRIAL: NCT04608591
Title: A Prospective Multicentre Study to Assess the Risk Factors That Contribute to Thrombosis in Patients With Lower Limb Injuries (R)Requiring Immobilisation to Identify High Risk Patients Requiring Thromboprophylaxis.
Brief Title: A Prospective Study to Assess the Risk Factors That Contribute to Thrombosis in Patients With Lower Limb Injuries.
Acronym: TILLIRI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Limerick (Other)
Responsible Party: Principal Investigator, Denis O'Keeffe, Consultant Haematologist, University of Limerick
Other Study IDs: TILLIRI
Record Dates: First submitted 2020-10-19; First posted 2020-10-29 (Actual); Last update posted 2020-10-29 (Actual); Status verified 2020-10

CONDITIONS: Thromboses, Venous; Lower Limb Injury
Keywords: Venous thromboembolism prophylaxis
MeSH Terms: conditions — Venous Thrombosis; Leg Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
* This study is aimed at identifying patients at high risk for Venous Thrombo-Embolism (VTE) (clots in the veins of legs or clots in the lungs) who have lower limb injuries treated with immobilisation of the lower limb. The study aims to identify high risk patients, who may benefit from thromboprophylaxis (blood thinning medication) to prevent such clots forming.
* To do this we will collect data on 3500 patients who present with lower limb injury requiring immobilisation to the Emergency Departments of the six hospitals named.
* We will assess their risk factors for venous thrombosis at the time of presentation and contact them at twelve weeks to assess if they have had a VTE in order to develop a risk scoring system which can be used to predict the likelihood of VTE development
* This risk scoring system can then be used to identify high risk patients who may benefit from thromboprophylaxis.

DETAILED DESCRIPTION:
Currently, there is wide variation in the provision of venous thromboembolism (VTE) prophylaxis for patients who suffer lower limb trauma and require lower limb immobilisation. Current United Kingdom guidelines recommend assessing competing risks of VTE and bleeding followed by shared decision-making with the patient on prescription of pharmacological thromboprophylaxis (VTE thromboprophylaxis). However, current American College of Chest Physicians (ACCP) guidelines do not recommend VTE thromboprophylaxis for this group. The largest study carried out to date, the Prevention of Thrombosis after Lower Leg Plaster Cast (POT-CAST) randomised controlled trial 1 identified a very low rate of VTE (1.8%) in the non-intervention arm. This study concluded that thromboprophylaxis was not justified for patients with lower limb trauma who required lower limb immobilisation. However, it recommended that further studies are required to see if it is possible to identify a high risk cohort of patients who may benefit from VTE thromboprophylaxis. No large prospective study has been published to date to assess if it is possible to identify this high risk group.

The Multiple Environmental and Genetic Assessment of risk factors for venous thrombosis (MEGA) study was a case-control study designed to identify risk factors for a first VTE. A sub-analysis of this study reviewed 230 patients who had lower limb trauma with cast immobilisation who developed VTE. Based on this data a risk assessment score was derived (termed "L-TRiP" [Leiden-Thrombosis Risk Prediction for patients with cast immobilization] score) in order to identify high risk patients who may benefit from VTE prophylaxis. However, this risk assessment tool has not been prospectively validated in a study.

We have carried out a pilot study to assess the feasibility of a large scale, adequately powered multi-centre study aimed at prospective identification of a high VTE-risk group of patients. This study was presented at the International Society on Thrombosis and Haemostasis meeting in Berlin in 2017.5 Utilizing data from this pilot study, we now aim to perform a multi-centre study with sufficient power to determine whether it is feasible to identify a high risk group of patients with lower limb trauma requiring immobilisation who will benefit from thromboprophylaxis The POT-CAST study determined that the rate of venous thrombo-embolism (VTE) in patients with lower limb trauma requiring a cast was 1.8%. This low rate does not justify VTE prophylaxis for all patients who require a cast. However there may be a high risk group with a rate of VTE high enough to suggest that consideration of VTE prophylaxis may be appropriate. This study will prospectively gather risk factor data on patients at the time of initial presentation post trauma with follow up at 12 weeks to identify those patients who have experienced a symptomatic VTE episode. This data will then be used to identify a group with a high VTE risk which future studies can utilise to target this high risk group to assess if VTE prophylaxis is of benefit.

ELIGIBILITY:
Inclusion Criteria:

* All patients who present to the Emergency Department with lower limb trauma requiring lower limb immobilisation. Aged over 18

Exclusion Criteria:

Patient unable to give consent Previous Venous thromboembolism

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients who present to the Emergency Departments of participating centres with lower limb injury over 18 requiring lower limb immobilisation.
Sampling Method: Probability Sample
Enrollment: 3500 (Estimated)
Dates: Start 2018-12-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
To measure the number of patients who develop venous thromboembolism within a 12 week period after a lower limb injury requiring immobilisation | 12 weeks post trauma and lower limb immobilisation
  All patients who present to the emergency department with lower limb injury ,require lower limb immobilisation and consent to the study will be enrolled in the study. At 12 weeks we will measure the number of patients who have developed a symptomatic venous thromboembolism confirmed by scanning to measure the rate of VTE in this population group.
The identification and measurement of the risk factors that contribute to the development of venous thromboembolism in patients with lower limb injury requiring immobilisation | 12 weeks post trauma and immobilisation
  To record in each participant individual thrombosis risk factors based on the Multiple Environmental and Genetic Assessment of risk factors for venous thrombosis study ( MEGA study) . To identify which of these factors are significantly associated with the development of venous thromboembolism in this population group.

SECONDARY OUTCOMES:
To identify a high risk group that will benefit from chemical prophylaxis | 12 weeks post trauma and immobilisation
  To combine the individual measured risk factors to develop a score that will identify a group of participants who are at high risk of thrombosis and will benefit from chemical prophylaxis

CONTACTS AND LOCATIONS:
Overall Officials: denis okeeffe, MBBCH, Principal Investigator — University of Limerick
Locations (1):
- Denis OKeeffe, Limerick, Ireland

IPD SHARING:
Plan to Share IPD: Yes
All researchers will input their centre patient data. The overall committee will review all patient data for review purposes . Individual centres will not be able to access other centres data.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: At the end of trial for a limited time.
Access Criteria: Only the reviewing committee will have access to all data. Individual centres will have access to their centres data.

REFERENCES:
- [Background] van Adrichem RA, Nemeth B, Algra A, le Cessie S, Rosendaal FR, Schipper IB, Nelissen RGHH, Cannegieter SC; POT-KAST and POT-CAST Group. Thromboprophylaxis after Knee Arthroscopy and Lower-Leg Casting. N Engl J Med. 2017 Feb 9;376(6):515-525. doi: 10.1056/NEJMoa1613303. Epub 2016 Dec 3. PMID 27959702
- [Background] Guyatt GH, Akl EA, Crowther M, Schunemann HJ, Gutterman DD, Lewis SZ. Introduction to the ninth edition: Antithrombotic Therapy and Prevention of Thrombosis, 9th ed: American College of Chest Physicians Evidence-Based Clinical Practice Guidelines. Chest. 2012 Feb;141(2 Suppl):48S-52S. doi: 10.1378/chest.11-2286. PMID 22315255
- [Background] Nemeth B, van Adrichem RA, van Hylckama Vlieg A, Bucciarelli P, Martinelli I, Baglin T, Rosendaal FR, le Cessie S, Cannegieter SC. Venous Thrombosis Risk after Cast Immobilization of the Lower Extremity: Derivation and Validation of a Clinical Prediction Score, L-TRiP(cast), in Three Population-Based Case-Control Studies. PLoS Med. 2015 Nov 10;12(11):e1001899; discussion e1001899. doi: 10.1371/journal.pmed.1001899. eCollection 2015 Nov. PMID 26554832
- [Background] Ocak G, Vossen CY, Verduijn M, Dekker FW, Rosendaal FR, Cannegieter SC, Lijfering WM. Risk of venous thrombosis in patients with major illnesses: results from the MEGA study. J Thromb Haemost. 2013 Jan;11(1):116-23. doi: 10.1111/jth.12043. PMID 23106832